CLINICAL TRIAL: NCT04644822
Title: A Phase 3, Non-randomized, Open Label, Multi-centre Clinical Trial to Investigate the Safety and Efficacy of [18F]PSMA-1007 Injection in Men With Suspected Persistent or Recurrent Prostate Cancer.
Brief Title: Safety and Efficacy of [18F]PSMA-1007 Injection in Suspected Persistent or Recurrent Prostate Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for Probe Development and Commercialization (Other)
Collaborators: McDougall Scientific Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CPD-002
Record Dates: First submitted 2020-11-11; First posted 2020-11-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer Recurrent; Recurrent Prostate Cancer
Keywords: prostate cancer; recurrent prostate cancer; persistent prostate cancer; PSMA; PET/CT; [18F]PSMA-1007
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]PSMA-1007 Injection (Experimental): A single dose of 3 - 4 MBq/kg Body Weight (up to a maximum of 400 MBq) of [18F]PSMA-1007 Injection will be administered followed by PET/CT imaging. (Patients on ADT treatment will receive the second dose approximately 6 months after the first dose)
  Interventions: Diagnostic Test: [18F] PSMA-1007 Injection

INTERVENTIONS:
Diagnostic Test: [18F] PSMA-1007 Injection — a novel [18F] PSMA radiotracer that is highly selective for PSMA.

SUMMARY:
This is a prospective, Phase 3 non-randomized, open label, multi-centre clinical trial to assess the safety and efficacy of [18F]PSMA-1007 Injection (investigational product or IP) in evaluating men with suspected persistent or recurrent disease (i.e., with biochemical failure), but with negative or equivocal conventional re-staging imaging (bone scan [BS] and computed tomography [CT] of abdomen and pelvis).

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and speak in English and provide informed consent
2. Male, Age ≥ 18 years
3. Prior primary treatment for prostate cancer with curative intent such as radical prostatectomy or radiotherapy for localized prostate cancer or other local or focal ablative therapy of the prostate
4. Not currently on systemic therapy (adjuvant or salvage) including androgen deprivation therapy
5. Suspected progressive or persistent disease after primary treatment for prostate cancer and biochemical failure (BF) with current management according to the following:

   1. Following primary radical prostatectomy (with or without adjuvant or salvage radiotherapy to the prostate bed/pelvis), where BF is defined as rising PSA on at least 2 occasions measured at least 1 month apart and with the most recent PSA measured within 3 months prior to enrollment at > 0.1 ng/mL
   2. Following primary radiotherapy (with either brachytherapy, external beam radiotherapy or combined brachytherapy and radiotherapy) for localized disease, where BF is defined according to the Phoenix Definition, which is rising PSA on at least 2 occasions measured at least 1 month apart and with the most recent PSA measured within 3 months prior to enrollment greater than the nadir PSA + 2.0 ng/mL
   3. Following primary ablative therapy to the prostate given with radical intent such as prior HIFU (high intensity focused ultrasound) or cryotherapy or other ablative energy therapy with biochemical failure as defined by the Stuttgart Criteria (nadir PSA + 1.2 ng/mL within 3 months prior to enrollment )
6. If PSA > 10 ng/mL, conventional imaging consisting of bone scan and CT scan within 3 months prior to consent that is either negative or equivocal.
7. Male subjects must be either:

   1. Documented by medical records or physician's note to be surgically sterile or,
   2. If capable of fathering a child, commit to the use of a barrier method of contraception, or agree to remain abstinent for 48 hours post-administration of the IP
8. Male subjects must agree to not donate sperm for 48 hours post-administration of the IP
9. Willing to participate in the study, is expected to be compliant, able to cooperate with study procedures, and have a high probability of completing the study in the opinion of the investigator
10. Vital sign results at Visit 1 and (pre-IP administration) at Visit 2 are within normal ranges, or if outside the normal ranges the results are judged by the investigator to not be clinically significant
11. Karnofsky performance status 70 or better (ECOG 0, 1)
12. Life expectancy of 6 months or more as judged by the investigator
13. Patient is medically suitable for salvage therapies

Exclusion Criteria:

1. Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components
2. Prior PSMA PET scan within 6 months of enrolment
3. Use of any other investigational medication or devices within 30 days prior to Visit 1
4. Known allergies or sensitivity to any component of the investigational product used in this study
5. Received significant ionizing radiation exposure, as judged by the Investigator, including from diagnostic or therapeutic radiopharmaceuticals used in clinical trials or for routine medical examinations, in the last 12 months
6. Undergoing ongoing occupational monitoring for radiation exposure
7. Clinically active, unstable, serious, life-threatening medical condition or disease that is, in the opinion of the Investigator, inadequately treated and/or where study participation may compromise the clinical management of the subject, or any other reason that makes the subject unsuitable to participate in this study
8. The participant has a history of alcohol or substance abuse
9. Patient cannot lie still for at least 30 minutes or comply with imaging procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: | 8 months
  • Imaging concordance (sensitivity, specificity, PPV, NPV) will be calculated by comparing presence or absence of disease based on PSMA-PET (at the patient level) compared with clinical outcome information (e.g., conventional imaging, clinical outcome surrogate or histopathologic correlate)

SECONDARY OUTCOMES:
Safety: Occurrence of AEs, SAEs, and changes from baseline in vital signs | 2 days
Percentage of patients identified with recurrent disease using [18F]PSMA-1007 | 2 months
Frequency with which [18F]PSMA-1007 PET/CT results lead to a change in recommended management | 2 months

OTHER OUTCOMES:
Percentage of patients with detectable disease relative to PSA levels | 2 months
Imaging concordance (sensitivity, specificity, PPV, NPV) based on [18F]PSMA-1007 PET/CT (at the regional level) compared with clinical outcome information (e.g., conventional imaging, clinical outcome surrogate or histopathologic correlate) | 8 months

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No